CLINICAL TRIAL: NCT02613377
Title: Transfusion-related Acute Lung Injury: a Prospective Cohort Study in Critically Ill Children
Acronym: TRALI
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Blood Services (Other)
Responsible Party: Principal Investigator, Dr Guillaume Emeriaud, MD, PhD, St. Justine's Hospital
Other Study IDs: CHUSJ-MP-21-2016-1070
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Acute Lung Injury
Keywords: Transfusion-related acute lung injury, Red Blood Cell
MeSH Terms: conditions — Acute Lung Injury; Transfusion-Related Acute Lung Injury | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — Blood samples will be collected from patients with suspected TRALI in order to generate some hypotheses regarding underlying mechanisms associated with the different types of TRALI (objective #2.e), the plasma level of IL-1beta, IL-6, IL8, and IL-10 will be measured.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Transfused critically ill children: Any infusion of RBC, plasma or platelets will be considered a transfusion.
  Interventions: Other: Blood transfusion
- Non-transfused critically ill children: For each transfused patient (index patient), one matched non-transfused control will be identified and included in the control group. The matching will be conducted using four criteria in hierarchical order: gender; age ± 10%; baseline Hemoglobin level (± 15 g/L); and Pediatric Risk of Mortality III score (PRISM III score ± 10%).

INTERVENTIONS:
Other: Blood transfusion
  Groups: Transfused critically ill children

SUMMARY:
Transfusions cause more adverse events in children than in adults. Patients in pediatric intensive care units (PICU) are particularly exposed to transfusions of plasma-rich blood products (red blood cell (RBC), plasma and platelets) and the risk of adverse events after a transfusion is particularly high in this vulnerable population. Transfusion-related acute lung injury (TRALI), an acute inflammation of the lungs that impairs gas exchange leading to acute respiratory failure, is one of the 2 most deadly transfusion complications in the general population. There is limited evidence on TRALI incidence and impact in critically ill children. This reduces the awareness of PICU team for this complication, and makes the decision process to transfuse particularly difficult. Moreover, acute lung injury is highly prevalent in critically ill children. It is therefore complex to ascertain if the high frequency of respiratory deteriorations observed after a transfusion in PICU is explained by the transfusion itself or by the evolution of the patient's critical illness.

The investigators will conduct a cohort study of consecutive transfused critically ill children, with a control group of matched non-transfused children. The primary objective is to determine if transfusion of RBC, plasma and/or platelets in PICU is an independent risk factor of TRALI, and to compare the respiratory evolution in the two matched (transfused and non-transfused) groups. The secondary objectives will include the determination of the incidence rate, risk factors and clinical impact of TRALI in transfused PICU patients. The investigators will study both "classic TRALI" and "delayed TRALI".

DETAILED DESCRIPTION:
Study Design This prospective cohort study will include all consecutive transfused patients admitted to the participating PICUs over a one-year period and a control group of matched non-transfused patients. The primary objectives will be assessed using the complete cohort of transfused and non-transfused patients. Secondary objectives will be studied in transfused patients.

Outcomes The primary outcome measure is TRALI (definite, probable, and delayed TRALI) as defined in section. In the non-transfused patients, the definition of Acute Lung Injury will be the same as the one used as a criterion for defining TRALI, and the observation period will be a similar 72-h period, starting at the same time zero.

Primary Objectives

* Objective #1a: to determine if the transfusion of RBC, plasma or platelets is an independent risk factor of TRALI in critically ill children.
* Objective #1b: to compare the progression of the respiratory function, in particular the SpO2/FiO2 ratio, in transfused and non-transfused PICU patients.

Secondary Objectives

* Objective #2.a : To determine the incidence rate of classic (definite or probable) TRALI and of delayed TRALI in transfused PICU patients.
* Objective #2.b : To characterize the risk factors of classic (definite or probable) TRALI and of delayed TRALI in transfused PICU patients.
* Objective #2.c : To compare the progression of respiratory parameters after a 1st transfusion in PICU patients with classic TRALI, delayed TRALI, and without TRALI.
* Objective #2.d : To compare the outcomes of transfused PICU patients with and without classic (definite or probable) TRALI and delayed TRALI.
* Objective #2.e : To describe the inflammatory profile of PICU patients with definite, probable, and delayed TRALI.

ELIGIBILITY:
Inclusion Criteria:

* admission to the PICU

Exclusion Criteria:

* gestational age < 40 weeks at entry into PICU
* post-term age less than 3 days or more than 18 years at PICU admission
* patients on extra-corporeal membrane oxygenation or ventricular assist device
* pregnancy present at entry into the PICU
* admission to PICU just after labor

Ages: 3 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children admitted to a participating PICU will be considered eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 717 (Actual)
Dates: Start 2016-01; Primary Completion 2020-01 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Transfusion-related acute lung injury | 72 hours

SECONDARY OUTCOMES:
Length of PICU stay (days) | 28 days
28-day all cause mortality | 28 days
Multiple organ dysfunction syndrome (MODS) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Emeriaud, MD, PhD, Principal Investigator — St. Justine's Hospital
Locations (4):
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - St. Justine's Hospital, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec